CLINICAL TRIAL: NCT01846507
Title: Tranexamic Acid in Adolescents With Heavy Menstrual Bleeding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Sarah O'Brien, Director of Experimental Therapeutics, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCH12-00822
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-09

CONDITIONS: Heavy Menstrual Bleeding
Keywords: Heavy Menstrual Bleeding; HMB; Lysteda
MeSH Terms: conditions — Menorrhagia | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tranexamic acid (Experimental): Subjects will complete a baseline menses (no treatment) followed by 3 menses using tranexamic acid.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Subjects will be instructed to take 2 tablets (1300) mg of Lysteda three times daily (3900 mg/daily) for five days during monthly menstruation.
  Other Names: Lysteda

SUMMARY:
This is a study to learn more about a drug called Tranexamic acid (TA), otherwise known as Lysteda, and whether or not this drug can decrease menstrual blood loss in young women and lead to an increase in the quality of life.

Menorrhagia in young women with bleeding disorders is typically treated with a combination of treatments including hormonal contraceptives. However, there are barriers to hormonal contraception use in younger adolescents.

Tranexamic acid is taken orally during the first 5 days of menstrual bleeding.

The purposes of this study include:

To test the safety and efficacy of Lysteda in adolescent females. To learn how well Lysteda works in decreasing menstrual blood loss. To see if parents and children participating in this study think the drug is improving their quality of life.

Lysteda has been approved by the Food and Drug Administration for use in patients > than 18 years of age but not for younger patients.

DETAILED DESCRIPTION:
This is a multi-center (5 sites) open-label, single-arm, efficacy study of Lysteda in the treatment of adolescent females (10-19 years of age) with heavy menstrual bleeding (HMB). Each subject will receive oral Lysteda 1.3 grams three times daily during the first five days of menses. Subjects will be monitored over the course of four menstrual cycles (1 pre-treatment cycle and 3 treatment cycles). During all cycles, assessments of menstrual bleeding will be performed using the Menorrhagia Impact Questionnaire (MIQ) and Pictorial Blood Assessment Chart (PBAC).

The study will begin as a currently funded pilot study to assess the efficacy of Lysteda in 32 patients followed to study completion.

ELIGIBILITY:
Inclusion Criteria:

1. Menstruating females 10-19 years of age
2. Non-smoker
3. Physician and patient have agreed to initiate Lysteda
4. Diagnosis of HMB based on the medical judgment of the principal or site investigator
5. Subjects must report menstrual periods occurring within 21-60 days from the start of one period to the start of the next menstrual period
6. Negative pregnancy test
7. Informed consent obtained and signed
8. Informed assent obtained and signed
9. Understanding of study procedures
10. Ability to comply with study procedures for the entire length of the study
11. Subjects should be either sexually inactive (abstinent) or agree to use a barrier method with spermicide in the event of sexual activity throughout the study period

Exclusion Criteria:

1. Active thromboembolic disease, history of thromboembolic disease (including retinal vein or artery occlusion), known inherited thrombophilia, or family history of thrombosis in a first degree relative
2. Subject has a severe medical or psychiatric illness that, in the opinion of the Investigator, would affect subject safety or compliance
3. Clinical evidence of severe bleeding disorder. Patients with mild bleeding disorders such as type 1 von Willebrand disease, mild platelet function defects such as platelet storage pool or release defects, and patients with bleeding due to Ehlers Danlos syndrome WILL be eligible to participate in the study.
4. Pregnancy within the past 6 months and/or breast-feeding
5. Use of hormonal contraception (estrogen and progestin) within 3 months of study entry, or anticipated need to initiate estrogen-containing hormonal contraception during the study period
6. Use of systemic steroids within 1 month of study entry
7. History of subarachnoid hemorrhage
8. History of Hepatitis B, C, or HIV
9. Baseline creatinine >20% above the upper limit of normal for age
10. Severe anemia (hemoglobin <8 g/dL)
11. Systolic blood pressure <85 or diastolic blood pressure <55
12. Heart rate <50 at time of screening
13. Use of intranasal DDAVP during menses will be permitted, but only if the patient has a history of using DDAVP consistently for ≥3 menstrual cycles prior to study enrollment, so that change in menstrual blood loss due to addition of Lysteda can be assessed. Use of one-time DDAVP during a DDAVP/Stimate challenge is also permitted during the study period, as is use of DDAVP in the event of severe epistaxis, trauma, or surgical procedures during the study period.

Ages: 10 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2013-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah O'Brien, MD, MSc, Principal Investigator — Nationwide Children's Hospital
Locations (5):
- United States (5):
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - Children's Mercy Hospital, Kansas City, Missouri
  - Akron Children's Hospital, Akron, Ohio
  - Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Baseline menses (no treatment) followed by 3 menses using tranexamic acid.
Groups:
- Tranexamic Acid: Adolescent girls aged 10-19 years with heavy menstrual bleeding
Period: Overall Study
Arm/Group | Tranexamic Acid
Started | 32
Completed | 25
Not Completed | 7
Not completed — Lost to Follow-up | 4
Not completed — Protocol Violation | 1
Not completed — Missing data | 2

BASELINE CHARACTERISTICS:
Arm/Group | Tranexamic Acid
Number analyzed (Participants) | 25
Age, Continuous [Mean (Full Range); unit: years] | 14.7 [11 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 14
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Menses for Participant Perceived Blood Loss
Description: Menorrhagia Impact Questionnaire (MIQ): Question 1 - participant perceived blood loss during most recent menses. Scale ranges from a score of 1 to 4 (with 1 being light blood loss and 4 being very heavy blood loss). Lower values indicate a better outcome (less blood loss during menses). Unit of measure is scores on a scale.
Time Frame: Baseline menses (no treatment) and 3 menstrual cycles treated with tranexamic acid
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Baseline Menses: Adolescent girls aged 10-19 with heavy menstrual bleeding - Baseline menses with no treatment
- Treated With Tranexamic Acid During Menses: Adolescent girls aged 10-19 years with heavy menstrual bleeding - treatment with Tranexamic Acid for 3 menses
Arm/Group | Baseline Menses | Treated With Tranexamic Acid During Menses
Number analyzed (Participants) | 25 | 25
score on a scale | 3 [1 to 4] | 1.9 [1 to 4]

2. Secondary Outcome: Change From Baseline Menses for Participant Perceived Limitation of School Attendance
Description: Menorrhagia Impact Questionnaire (MIQ): Question 2 - participant perceived limitation of school attendance during most recent menses. Scale ranges from a score of 1 to 5 (with 1 being school attendance not at all limited and 5 being school attendance limited extremely). Lower values indicate a better outcome (less limitation of school attendance). Unit of measure is scores on a scale.
Time Frame: Baseline menses (no treatment) and 3 menstrual cycles treated with tranexamic acid
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Baseline Menses: Adolescent girls aged 10-19 years with heavy menstrual bleeding - Baseline menses with no treatment
Arm/Group | Baseline Menses | Treated With Tranexamic Acid During Menses
Number analyzed (Participants) | 25 | 25
score on a scale | 1.64 [1 to 5] | 1.27 [1 to 5]

3. Secondary Outcome: Change From Baseline Menses for Participant Perceived Limitation in Physical Activities
Description: Menorrhagia Impact Questionnaire (MIQ): Question 3 - participant perceived limitation in physical activities during most recent menses. Scale ranges from a score of 1 to 5 (with 1 being physical activities not at all limited and 5 being physical activities extremely limited). Lower values indicate a better outcome (less limitation of physical activities). Unit of measure is scores on a scale.
Time Frame: Baseline menses (no treatment) and 3 menstrual cycles treated with tranexamic acid
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Baseline Menses | Treated With Tranexamic Acid During Menses
Number analyzed (Participants) | 25 | 25
score on a scale | 2.08 [1 to 5] | 1.40 [1 to 5]

4. Secondary Outcome: Change From Baseline Menses for Participant Perceived Limitation of Social or Leisure Activities
Description: Menorrhagia Impact Questionnaire (MIQ): Question 4 - participant perceived limitation of social or leisure during most recent menses. Scale ranges from a score of 1 to 5 (with 1 being social or leisure activities not at all limited and 5 being social or leisure activities limited extremely). Lower values indicate a better outcome (less limitation of social or leisure activities). Unit of measure is scores on a scale.
Time Frame: Baseline menses (no treatment) and 3 menstrual cycles treated with tranexamic acid
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Baseline Menses | Treated With Tranexamic Acid During Menses
Number analyzed (Participants) | 25 | 25
score on a scale | 3.5 [1 to 5] | 1.76 [1 to 5]

5. Secondary Outcome: Change From Baseline Menses for Menstrual Blood Loss as Measured by Pictorial Blood Assessment Chart (PBAC) Scores
Description: Pictorial Blood Assessment Chart (PBAC) scores - participant assessment of menstrual blood loss during menses using a pictorial chart to score menstrual blood loss. Pictorial scores range from 1 point for mild soaking of a pad/tampon, 5 points for moderate soaking of a pad/tampon, 10 points for severe soaking of a pad/tampon, and 5 points for each episode of flooding and for each blood clot larger than a quarter in size. Lower values indicate a better outcome (less blood loss). Unit of measure is a total computed score (all points during the menses from the pictorial chart added together).
Time Frame: Baseline menses (no treatment) and 3 menstrual cycles treated with tranexamic acid
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Baseline Menses | Treated With Tranexamic Acid During Menses
Number analyzed (Participants) | 24 | 24
score on a scale | 255.1 [62 to 699] | 154.6 [12 to 561]

6. Secondary Outcome: Change From Baseline Menses for Hemoglobin Lab Value
Description: Hemoglobin lab value normal range is 12 g/dL to 16 g/dL. Values in the range of 12 g/dL to 16 g/dL would be considered normal Hemoglobin values. A score lower than the normal range (below 12 g/dL) would indicate a worse outcome. Unit of measure is g/dL.
Time Frame: Baseline menses (no treatment) and 3 menstrual cycles treated with tranexamic acid
Measure: Mean (Full Range); unit: gm/dL
Arm/Group | Baseline Menses | Treated With Tranexamic Acid During Menses
Number analyzed (Participants) | 25 | 22
gm/dL | 12.67 [10.4 to 15.3] | 12.84 [10.6 to 14.7]

7. Secondary Outcome: Change From Baseline Menses for Ferritin Lab Value
Description: Ferritin lab value normal range is 7 ng/mL to 142 ng/mL. Values in the range of 7ng/mL to 142 ng/mL would be considered normal Ferritin values. A score lower than the normal range (below 7 ng/mL) would indicate a worse outcome. Unit of measure is ng/mL.
Time Frame: Baseline menses (no treatment) and 3 menstrual cycles treated with tranexamic acid
Measure: Mean (Full Range); unit: ng/dL
Arm/Group | Baseline Menses | Treated With Tranexamic Acid During Menses
Number analyzed (Participants) | 25 | 22
ng/dL | 25.94 [4 to 82] | 26.34 [5 to 59]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Tranexamic Acid
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 23/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranexamic Acid (N=30)
Suicidal Ideation (Psychiatric disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranexamic Acid (N=30)
Fatigue (Reproductive system and breast disorders) | 6 (8)
Headache (General disorders) | 5 (7)
Upper respiratory infection sypmtoms (Infections and infestations) | 14 (23)
Dysmenorrhea (Reproductive system and breast disorders) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 (10)
Abdominal pain (Gastrointestinal disorders) | 6 (7)
Heavy menses (Reproductive system and breast disorders) | 2 (3)
Anxiety (Psychiatric disorders) | 2 (2)
Fever (Infections and infestations) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (4)
Dizziness (General disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Small sample size Subjective measurement of menstrual blood loss

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No